CLINICAL TRIAL: NCT04812457
Title: Effectiveness of Hyaluronic Acid in Postoperative Cures in Partial Matriceptomes With the Phenol/Alcohol Technique. Randomized Clinical Trial
Brief Title: Hyaluronic Acid in Postoperative Cures in the Phenol/Alcohol Technique
Acronym: EHAPAT
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Gabriel Gijon-Nogueron, Associate Professor, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UMalagaUEX2021
Record Dates: First submitted 2021-03-13; First posted 2021-03-23 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Nails, Ingrown; Hyaluronic Acid
Keywords: matriceptomies; wound; nail
MeSH Terms: conditions — Nails, Ingrown; Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physiological cures using pure hyaluronic acid (Hialucic®) (Experimental): After the intervention of unilateral onychocryptosis, the partial matricectomy technique with phenol / alcohol,next to an ointment with hyaluronic acid (hyalucic ®) will be used together with a non-stick dressing and a semi-compression bandage to prevent bleeding
  Interventions: Drug: Hialucic
- Control group using traditional cure (Betadine Gel). (Active Comparator): After the intervention of unilateral onychocryptosis, the partial matricectomy technique with phenol / alcohol,next to Povidone Iodine Gel (Betadine Gel®) will be applied following the same procedure.
  Interventions: Drug: Betadine gel

INTERVENTIONS:
Drug: Hialucic — A professional not present at the intervention (researcher 2) will proceed to carry out the postoperative cures 48 hours after the intervention. The bandage will be removed, the area will be washed with physiological saline and the drug will be applied according to the group to which it belongs. In the intervention group, an ointment with hyaluronic acid (hyalucic ®) will be used together with a non-stick dressing and a semi-compression bandage to prevent bleeding.
  Arms: Physiological cures using pure hyaluronic acid (Hialucic®)
Drug: Betadine gel — A professional not present at the intervention (researcher 2) will proceed to carry out the postoperative cures 48 hours after the intervention. The bandage will be removed, the area will be washed with physiological saline and the drug will be applied according to the group to which it belongs. In the control group, Betadine Gel will be used together with a non-stick dressing and a semi-compression bandage to prevent bleeding.
  Arms: Control group using traditional cure (Betadine Gel).

SUMMARY:
The purpose of this study is to compare the efficacy of a postoperative treatment protocol with hyaluronic acid-based ointment compared to the standard protocol (betadine gel) in partial chemical matricectomies with phenol alcohol technique. This will allow to see if the use of hyaluronic acid could help to reduce the healing time and total recovery of this surgical technique

DETAILED DESCRIPTION:
A randomized controlled multicenter study will be conducted. Subject (n=60) will be adolescent and healthy adults, between 14 and 40 years old, who require and demand surgical treatment of onychocryptosis or stage I or IIa ingrown nail in the participating centers.

After acceptance to participate in the study, they will be operated on in a standardized protocol with phenol-alcohol technique. Then they will be randomly assigned into 2 groups, to perform different treatment protocols. The experimental group will receive physiological cures using pure hyaluronic acid (Hialucic®) after the onychocryptosis surgery, while the control group will receive traditional cure (Betadine Gel). The periodicity of cures in both groups will be the same, 48 hours, 6 days, 12 days 16 days and 20 days. For the design of the study, the bases on randomized clinical studies described in CONSORT will be followed.

The outcome measurement will be the presence of exudate in each of the cures (carried out at the same post-surgical times), presence or absence of granulation tissue, reduction of inflammation (measured with the circumference of the finger in the eponychium area), cost average treatment protocol, time elapsed until primary healing (when the wound stops staining the bandage) and final surgical discharge (finger without wound or inflammation), referred pain in the finger during the healing period and presence of complications, such like persistent inflammation, infection, etc.

PARTICIPANTS

Participants will be recruited through the Podiatric Clinic of the University of Extremadura and Lopezosa y Gijon Nogueron clinics in Malaga and Granada

SAMPLE´S SIZE CALCULATION

The confidence level was established at 95% and the statistical power at 90%. We need a minimum precision value of 3 days (time between cures). The squared variance (S2) is 16, since in a previous pilot study the variance between groups of cures was 4 days

The inclusion criteria were as follows:

* Patients aged between 14 and 40 years old
* Patients with stage I, II, or III onychocryptosis (Kline classification) or Mozena stage I or IIa [7]
* Patients with onychocryptosis unilateral or bilateral.
* Healthy patients without previous systematic pathologies (diabetes, coagulation or immunological disorders) who require and demand surgical treatment of their pathology in the participating centers and willing to participate in the study.

Participants were excluded if any of the following were present:

* Onychocyptosis with significant involvement of the hypertrophic labrum
* Patients with hyperhidrosis
* Severe paronychias
* Allergy to any of the substances used in the intervention or in the cures.

2.3 RANDOMIZATION Participants will be divided into two groups: a) experimental or intervention group (hyaluronic acid cures) and b) control group (Betadine Gel cures) by random assignment of sealed envelopes, which will be previously sealed in sequential order. Both the patient and the researcher will be blinded to hide the group to which each patient belongs.

2.4 INTERVENTION

For the intervention of unilateral onychocryptosis, the partial matricectomy technique with phenol / alcohol will be carried out. After removal of the affected spicule, basic manual curettage will be performed with a Wolkmann or Martini spoon. Once the matrix has been mechanically removed, the phenol will be applied. Phenol 88% in sterile capsules will be used in the affected canal using a cotton swab for two applications of 30 seconds. Between these two applications, alcohol will be used to dissolve the phenol present in the nail bed. After the last application of phenol, the area will be washed again with alcohol.

After the intervention, hyaluronic acid will be applied in the operated canal. A non-stick dressing impregnated with Betadine will be placed and a semi-compression bandage will be applied.

A professional not present at the intervention (researcher 2) will proceed to carry out the postoperative cures 48 hours after the intervention. The bandage will be removed, the area will be washed with physiological saline and the drug will be applied according to the group to which it belongs. In the intervention group, an ointment with hyaluronic acid (hyalucic ®) will be used together with a non-stick dressing and a semi-compression bandage to prevent bleeding. In the control group, Povidone Iodine Gel (Betadine Gel®) will be applied following the same procedure.

Successive cures will be carried out every 2 days by the healthcare professional, where both groups will be washed with saline solution and a new dose of ointment will be applied as appropriate in each group. hyaluronic acid for cures a maximum of 4 times, to avoid maceration of the wound. the rest of the cures will be with Betadine. Primary healing will be taken as the first variable of surgical results and the definitive discharge time, which will be determined by researcher 2 (who was responsible for the cures) and confirmed by a third evaluator, who will verify the results.

2.5 OUTCOME MEASURE

The demographic characteristics of the participants will be age, sex, and onychocryptosis classification according to Kline or Mozena.

The variables to be used are:

* Dressing application time (time recorded in min).
* Presence of exudate (Very Abundant / Abundant / Slight / Absent).
* Reduction of inflammation, measured in mm with flexible tape around the eponychium.
* Cost (average costs for all materials used per patient in €),
* Visual analog scale pain (VAS)
* Presence of complications such as infection (noted at the end of treatment or dressing change).
* Time elapsed until the primary healing and total healing of the wound (days).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 14 and 40 years old
* Patients with stage I, II, or III onychocryptosis (Kline classification) or Mozena stage I or IIa
* Patients with onychocryptosis unilateral or bilateral.
* Healthy patients without previous systematic pathologies (diabetes, coagulation or immunological disorders) who require and demand surgical treatment of their pathology in the participating centers and willing to participate in the study.

Exclusion Criteria:

* Onychocyptosis with significant involvement of the hypertrophic labrum
* Severe paronychias
* Allergy to any of the substances used in the intervention or in the cures.

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2021-03-06 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Time elapsed until the primary healing and total healing of the wound | from the intervention until 15 weeks late
  We measure the days that the patients wait to see the wound perfectly between 0 days until 300 days

SECONDARY OUTCOMES:
Presence of exudate | from the intervention until 15 weeks late
  (Very Abundant / Abundant / Slight / Absent).
Reduction of inflammation | from the intervention until 15 weeks late
  measured in mm with flexible tape around the eponychium
cost | from the intervention until 15 weeks late
  average costs for all materials used per patient in €
Visual analog scale pain | from the intervention until 15 weeks late
  Visual analog scale pain between 0 to 100 mm
Presence of complications such as infection | from the intervention until 15 weeks late
  Noted at the end of treatment or dressing change

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Gijon-Nogueron, PhD, Principal Investigator — University of Malaga
Locations (1):
- Eva Lopezosa Reca, Málaga, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andreassi A, Grimaldi L, D'Aniello C, Pianigiani E, Bilenchi R. Segmental phenolization for the treatment of ingrowing toenails: a review of 6 years experience. J Dermatolog Treat. 2004 Jun;15(3):179-81. doi: 10.1080/09546630410026860. PMID 15204151
- [Background] Hassel JC, Hassel AJ, Loser C. Phenol chemical matricectomy is less painful, with shorter recovery times but higher recurrence rates, than surgical matricectomy: a patient's view. Dermatol Surg. 2010 Aug;36(8):1294-9. doi: 10.1111/j.1524-4725.2010.01625.x. Epub 2010 Jun 22. PMID 20573174
- [Background] Giacalone VF. Phenol matricectomy in patients with diabetes. J Foot Ankle Surg. 1997 Jul-Aug;36(4):264-7; discussion 328. doi: 10.1016/s1067-2516(97)80070-1. PMID 9298440
- [Background] Karaca N, Dereli T. Treatment of ingrown toenail with proximolateral matrix partial excision and matrix phenolization. Ann Fam Med. 2012 Nov-Dec;10(6):556-9. doi: 10.1370/afm.1406. PMID 23149533